CLINICAL TRIAL: NCT04210245
Title: Evaluation of Efficacy, Safety and Tolerability of NGM282 (Aldafermin) in a Phase 2b, Randomized, Double-blind, Placebo-controlled, Multi-center Study in Subjects With Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis (ALPINE 4)
Brief Title: Study of Aldafermin (NGM282) in Subjects With Compensated Cirrhosis (ALPINE 4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 282-CC-207
Record Dates: First submitted 2019-12-16; First posted 2019-12-24 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Compensated Cirrhosis; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Daily 0.3 mg dose (Experimental): Administered by subcutaneous injection
  Interventions: Biological: aldafermin
- Daily 1 mg dose (Experimental): Administered by subcutaneous injection
  Interventions: Biological: aldafermin
- Daily 3 mg dose (Experimental): Administered by subcutaneous injection
  Interventions: Biological: aldafermin
- Placebo (Placebo Comparator): Administered by subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: aldafermin — aldafermin
  Arms: Daily 0.3 mg dose; Daily 1 mg dose; Daily 3 mg dose
Other: Placebo — Placebo for aldafermin
  Arms: Placebo

SUMMARY:
A multi-center evaluation of aldafermin in a randomized, double-blind, placebo-controlled study in subjects with compensated cirrhosis.

DETAILED DESCRIPTION:
The study will compare multiple doses of aldafermin against placebo in a compensated NASH cirrhosis population for 48 weeks of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Liver biopsy consistent with NASH cirrhosis.
2. Compensated cirrhosis due to NASH.

Key Exclusion Criteria:

1. Other causes of liver disease including but not limited to alcoholic liver disease, hepatitis B, hepatitis C, autoimmune disorders, primary biliary cirrhosis, drug-induced hepatotoxicity, Wilson's disease, hemochromatosis, and alpha-1-anti-trypsin definition based on medical history and/or centralized read of liver histology.
2. Evidence of drug induced steatohepatitis secondary to amiodarone, corticosteroids, estrogens, methotrexate, tetracycline, or other medications known to cause hepatic steatosis.
3. History of hepatic decompensation including variceal bleeding, ascites, or hepatic encephalopathy.
4. Model of end stage liver disease (MELD) score >12.

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals
Locations (43):
- United States (26):
  - NGM Clinical Study Site, Glendale, Arizona
  - NGM Clinical Study Site 413, Tucson, Arizona
  - NGM Clinical Study Site 415, Tucson, Arizona
  - NGM Clinical Study Site, North Little Rock, Arkansas
  - NGM Clinical Study Site, Fresno, California
  - NGM Clinical Study Site, La Jolla, California
  - NGM Clinical Study Site, Los Angeles, California
  - NGM Clinical Study Site, Panorama City, California
  - NGM Clinical Study Site, Rialto, California
  - NGM Clinical Study Site, Boca Raton, Florida
  - NGM Clinical Study Site, Miami, Florida
  - NGM Clinical Study Site, Marietta, Georgia
  - NGM Clinical Study Site, Chicago, Illinois
  - NGM Clinical Study Site, Baltimore, Maryland
  - NGM Clinical Study Site, Boston, Massachusetts
  - NGM Clinical Study Site, Flowood, Mississippi
  - NGM Clinical Study Site 488, Jackson, Mississippi
  - NGM Clinical Study Site, Kansas City, Missouri
  - NGM Clinical Study Site, Durham, North Carolina
  - NGM Clinical Study Site, Germantown, Tennessee
  - NGM Clinical Study Site, Austin, Texas
  - NGM Clinical Study Site, Edinburg, Texas
  - NGM Clinical Study Site 481, Houston, Texas
  - NGM Clinical Study Site, San Antonio, Texas
  - NGM Clinical Study Site, Richmond, Virginia
  - NGM Clinical Study Site 482, Seattle, Washington
- Australia (8):
  - NGM Clinical Study Site, Camperdown, New South Wales
  - NGM Clinical Study Site, Westmead, New South Wales
  - NGM Clinical Study Site, Adelaide, South Australia
  - NGM Clinical Study Site, Bedford Park, South Australia
  - NGM Clinical Study Site, Clayton, Victoria
  - NGM Clinical Study Site, Fitzroy, Victoria
  - NGM Clinical Study Site, Heidelberg, Victoria
  - NGM Clinical Study Site, Melbourne, Victoria
- NGM Clinical Study Site, Brussels, Belgium
- France (2):
  - NGM Clinical Study Site, Paris
  - NGM Clinical Study Site, Pessac
- NGM Clinical Study Site, Leipzig, Germany
- NGM Clinical Study Site, Shatin, Hong Kong
- Poland (2):
  - NGM Clinical Study Site 444, Wroclaw
  - NGM Clinical Study Site 446, Wroclaw
- NGM Clinical Study Site, San Juan, Puerto Rico
- NGM Clinical Study Site 466, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rinella ME, Lieu HD, Kowdley KV, Goodman ZD, Alkhouri N, Lawitz E, Ratziu V, Abdelmalek MF, Wong VW, Younes ZH, Sheikh AM, Brannan D, Freilich B, Membreno F, Sinclair M, Melchor-Khan L, Sanyal AJ, Ling L, Harrison SA. A randomized, double-blind, placebo-controlled trial of aldafermin in patients with NASH and compensated cirrhosis. Hepatology. 2024 Mar 1;79(3):674-689. doi: 10.1097/HEP.0000000000000607. Epub 2023 Sep 21. PMID 37732990

RESULTS

PARTICIPANT FLOW:
Groups:
- Daily 0.3 mg Dose; Daily 1 mg Dose; Daily 3 mg Dose; Placebo: Administered by subcutaneous injection daily for 48 weeks
Period: Overall Study
Arm/Group | Daily 0.3 mg Dose | Daily 1 mg Dose | Daily 3 mg Dose | Placebo
Started | 7 | 42 | 55 | 56
Completed | 7 | 37 | 44 | 49
Not Completed | 0 | 5 | 11 | 7
Not completed — Adverse Event | 0 | 3 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 4
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — 1 due to life stressors and injection site discomfort and 1 subject started prohibited medication | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily 0.3 mg Dose | Daily 1 mg Dose | Daily 3 mg Dose | Placebo | Total
Number analyzed (Participants) | 7 | 42 | 55 | 56 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 24 | 37 | 45 | 111
  >=65 years | 2 | 18 | 18 | 11 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.78) | 61.3 (7.57) | 59.6 (8.72) | 58.3 (8.11) | 59.6 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 23 | 36 | 39 | 103
  Male | 2 | 19 | 19 | 17 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 12 | 18 | 40
  Not Hispanic or Latino | 4 | 33 | 43 | 38 | 118
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 4 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 3
  White | 7 | 38 | 47 | 46 | 138
  More than one race | 0 | 2 | 1 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter] — centimeter
  centimeter | 164.3 (11.35) | 167.5 (11.23) | 166.2 (10.02) | 163.9 (8.89) | 165.7 (10.05)
Weight [Mean (Standard Deviation); unit: kilogram] — kilogram
  kilogram | 88.19 (9.680) | 101.47 (22.240) | 95.27 (22.407) | 93.43 (19.906) | 95.95 (21.255)
BMI [Mean (Standard Deviation); unit: kg/m^2] — kg/m^2
  kg/m^2 | 32.768 (3.2236) | 35.979 (6.3231) | 34.265 (6.7146) | 34.757 (7.1164) | 34.822 (6.6468)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Enhanced Liver Fibrosis Score at Week 48
Description: Enhanced Liver Fibrosis (ELF) score is a non-invasive blood test derived from the measurement of hyaluronic acid (HA), amino terminal propeptide of type III procollagen (PIIINP), and tissue inhibitor of metalloprotease 1 (TIMP1) using a proprietary algorithm (Siemens). ELF score is a laboratory test, is unitless, and is used as a continuous variable. The minimal ELF score is zero, the maximal ELF score is unknown. The higher the ELF score, the worse the disease outcome.
  ELF is a score on a scale of severity assessment against biopsy-proven fibrosis. A score of <7.7 is none to mild, > 7.7-9.8 is moderate, > 9.8 is severe.
Time Frame: 48 weeks
Population: Enrollment to the 0.3 mg dose treatment arm was terminated during the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily 0.3 mg Dose | Daily 1 mg Dose | Daily 3 mg Dose | Placebo
Number analyzed (Participants) | 7 | 37 | 44 | 49
score on a scale | -0.071 (0.7214) | 0.125 (0.6938) | -0.213 (0.6145) | 0.263 (0.5767)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from consenting to the end of study (1 years)
Arm/Group | Daily 0.3 mg Dose | Daily 1 mg Dose | Daily 3 mg Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/42 | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/7 | 11/42 | 5/55 | 3/56
Other Adverse Events (participants affected / at risk) | 5/7 | 40/42 | 52/55 | 49/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily 0.3 mg Dose (N=7) | Daily 1 mg Dose (N=42) | Daily 3 mg Dose (N=55) | Placebo (N=56)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily 0.3 mg Dose (N=7) | Daily 1 mg Dose (N=42) | Daily 3 mg Dose (N=55) | Placebo (N=56)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 6 (6) | 7 (7) | 5 (5)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Reaction to food additive (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 2 (2) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 4 (4) | 6 (6)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 8 (8) | 5 (5)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 | 0 (0) | 1 (1) | 3 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3) | 6 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (6) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 7 (7) | 10 (10)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5) | 8 (8) | 7 (7)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 12 (12) | 18 (18) | 5 (5)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5) | 3 (3)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (5) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 7 (7) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 14 (14) | 13 (13) | 17 (17)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 4 (4) | 9 (9)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 8 (8) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 11 (11) | 22 (22) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04210245/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT04210245/SAP_001.pdf